CLINICAL TRIAL: NCT05433883
Title: The Relationship Between Obstructive Sleep Apnea and Alzheimer's Disease: Evidence and Effectiveness
Acronym: OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hsueh-Yu Li
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea of Adult; Mild Cognitive Impairment
Keywords: Alzheimer's disease; Obstructive Sleep Apnea
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: The research plan to enroll 15 simple snoring patients (apnea/hypopnea <5, control group), 30 severe OSA patients (apnea/hypopnea >30, treatment group), and 15 mild cognitive impairment patients (comparative group). All patients complete Mini-Mental State Examination, peripheral blood sample for plasma Aβ42, Aβ40, Aβ42/Aβ40, Tau, NfL; amyloid deposit in18F-florbetapir PET; and Taiwan smell identification test. Thirty severe OSA patients (AHI>30, treatment group) receive comprehensive upper airway surgery with/without bariatric surgery and repeat postoperative assessment in polysomnography and aforementioned examinations 1 year later.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treatment group (Experimental): 30 severe OSA patients (apnea/hypopnea >30)
  Interventions: Procedure: sleep surgery
- control group (No Intervention): 15 simple snoring patients (apnea/hypopnea <5 )
- comparative group (No Intervention): 15 mild cognitive impairment patients.

INTERVENTIONS:
Procedure: sleep surgery — Thirty severe OSA patients (AHI>30, treatment group) receive comprehensive upper airway surgery with/without bariatric surgery and repeat postoperative assessment in polysomnography and aforementioned examinations 1 year later.
  Other Names: comprehensive upper airway surgery
  Arms: treatment group

SUMMARY:
The research plan to enroll 15 simple snoring patients (apnea/hypopnea <5, control group), 30 severe OSA patients (apnea/hypopnea >30, treatment group), and 15 mild cognitive impairment patients (comparative group). All patients complete Mini-Mental State Examination, peripheral blood sample for plasma Aβ42, Aβ40, Aβ42/Aβ40, Tau, NfL; amyloid deposit in18F-florbetapir PET; and Taiwan smell identification test. Thirty severe OSA patients (AHI>30, treatment group) receive comprehensive upper airway surgery with/without bariatric surgery and repeat postoperative assessment in polysomnography and aforementioned examinations 1 year later.

DETAILED DESCRIPTION:
Obstructive sleep apnea and Alzheimer's disease are both highly prevalent and age-related chronic disease with significant impacts on global public health. The link between OSA and AD showed an inter-dependent relationship. Our genetic study showed the expressions of AD-associated genes (CCL2, IL6, CXCL8, HLA-A, IL1RN) in severe OSA patients. Our epidemiological study revealed OSA patients were significantly associated with a higher incidence of AD (adjusted hazard ratio: 2.12) in comparison to non-OSA subjects and treated OSA patients exhibited a significantly reduced risk of AD (incidence rate ratio: 0.23) compared with non-treated OSA patients. Possible mechanisms of OSA in contributing to AD are sleep fragmentation, intermittent hypoxia, intrathoracic swings, and olfactory dysfunction. The cognitive decline in AD seems progressive and irreversible, by contrast, OSA sharing similar cognitive impairment is treatable. The purposes of this study are (1) to explore the relationship and mechanism between OSA and AD, and establish an alarm system as early stage of AD in OSA patients, (2) to testify the improvement of OSA can feedback to ameliorate cognitive impairment and modify the process of AD.

The research plan to enroll 15 simple snoring patients (apnea/hypopnea <5, control group), 30 severe OSA patients (apnea/hypopnea >30, treatment group), and 15 mild cognitive impairment patients (comparative group). All patients complete Mini-Mental State Examination, peripheral blood sample for plasma Aβ42, Aβ40, Aβ42/Aβ40, Tau, NfL; amyloid deposit in18F-florbetapir PET; and Taiwan smell identification test. Thirty severe OSA patients (AHI>30, treatment group) receive comprehensive upper airway surgery with/without bariatric surgery and repeat postoperative assessment in polysomnography and aforementioned examinations 1 year later.

The data from the study can be used to explore the association between polysomnography and AD-related examinations, to compare the perioperative changes in polysomnography and AD-related examinations, to correlate the perioperative changes between polysomnography and AD-related examinations. The contributions of the study are to clarify the hypothesis: severe OSA is early stage and one of the etiology contributing to the development of AD, and sleep surgery improves OSA and consequently modify the process of AD, early detection of cognition and olfactory function in OSA patients can contribute to diagnosis of early stage AD and consequently early treatment to modify the development of AD.

ELIGIBILITY:
Inclusion Criteria:

1. age >50 years
2. control group, AHI<5 (n=15)
3. treatment group, AHI>30 (n=30)
4. Comparative group, mild cognitive impairment (n=15)

Exclusion Criteria:

The exclusion criteria were definite neurologic disorders affecting brain structure (e.g., stroke, traumatic head injury or epilepsy), unstable medical diseases involving the heart, lungs, liver or kidneys, chronic insomnia, allergic rhinitis/paranasal sinusitis and alcohol or substance abuse/dependence currently or in the past one year.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
polysomnography | one year
  simple snoring patients (apnea/hypopnea <5),severe OSA patients (apnea/hypopnea >30)

SECONDARY OUTCOMES:
Mini-Mental State Examination | one year
  Cognitive assessment in the present study is Mini Mental Status Examination (MMSE). The MMSE is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
peripheral blood sample for plasma Aβ42, Aβ40, Aβ42/Aβ40, Tau, NfL | one year
  Every subject provided a 20-ml venous blood sample (K3 EDTA, lavender-top tube). Samples were collected under non-fasting conditions between 9 AM and 2 PM. The blood samples were centrifuged at 3,000 × g for 20 minutes within half an hour of collection, and then plasma was aliquoted into cryotubes (1 ml per tube) and stored at -80 °C.
amyloid deposit (18F-florbetapir PET) | one year
  The radiosynthesis of 18F-florbetapir (AV-45) and amyloid PET data acquisition followed the same procedures as previously described . A fixed dose approximate of 10mCi (370 MBq) 18F-florbetapir (AV-45) will be given to each subject. 10-minute image will be acquired 50-60min post injection using a Biograph mMR PET/MR System or PET/CT scanner.
Taiwan smell identification test | one year
  The TWSIT questionnaire consisted of two questionnaires (test 1 and test 2), which contained the same multi-choice questions but in different sequence. Eight odorants (honey, peach, passion fruit, cantaloupe, lemon, smoked plum, garlic, coffee, jasmine), which are familiar to Taiwanese with a high identification rate (more than 95%), were identified and used in the questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: professor, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan